CLINICAL TRIAL: NCT04629274
Title: IMCY-NMO-000 In Vitro Study of the Biological and Immunological Activity of Imotopes® Candidates on Blood Cells of Patients With Stabilized Neuromyelitis Optica (PHASE 0)
Brief Title: In Vitro Study of the Biological and Immunological Activity of Imotopes® Candidates on Blood Cells of Patients With Stabilized NMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imcyse SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IMCY-NMO-000
Record Dates: First submitted 2020-10-29; First posted 2020-11-16 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Neuromyelitis Optica
MeSH Terms: conditions — Neuromyelitis Optica | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test of Imotopes® candidates on blood cells of patients with stabilized NMO (Experimental): To test in vitro the binding of different Imotopes® to class II HLA antigens on PBMC isolated from patients presenting a diagnosed and stabilized neuromyelitis optica spectrum disorders, as well as their ability to generate a cytolytic response directed against the immune cells involved in the maintenance and triggering of the disease (i.e. non-cytolytic T cells recognising the same epitopes and antigen presenting cells (APC) presenting the same epitopes).
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — The patients will be asked to provide at least 2 peripheral blood samples of approximately 100 milliliters each time, with a minimum of 14 days interval between these 2 samples.If the results obtained with the 2 initial samples would be of interest to the Sponsor, the patient will be asked to come back for additional samplings with a maximum of 6 additional blood draws

SUMMARY:
This is a fundamental, prospective, multi-centres, interventional non-comparative study without the administration of a study product to patients.

A phase 0 study is particularly well adapted to early exploration of potential targeted treatments - i.e. treatments whose efficacy can only be hoped for in patients presenting specific biological characteristics in addition to being diagnosed with the targeted disease, Neuromyelitis Optica Spectrum Disorders (NMOSD) in this study. The main goal of the study will be to support the selection of Imotopes® (i.e. synthetic peptides encompassing HLA Class II T epitopes flanked by a thioreductase motif), and (i) capable of binding with class II HLA antigens of each patient and (ii) causing ex vivo the appearance of epitope -specific cytolytic CD4+ T cells.

DETAILED DESCRIPTION:
This is a fundamental, prospective, multi-centres, interventional non-comparative study without the administration of a study product to patients.

The objective is to test in vitro the binding of different Imotopes® to class II HLA antigens on peripheral blood mononuclear cell (PBMC) isolated from patients presenting a diagnosed and stabilized neuromyelitis optica spectrum disorders, as well as their ability to generate a cytolytic response directed against the immune cells involved in the maintenance and triggering of the disease (i.e. non-cytolytic T cells recognising the same epitopes and antigen presenting cells (APC) presenting the same epitopes).

The patients will be asked to provide at least 2 peripheral blood samples of approximately 100 milliliters each time, with a minimum of 14 days interval between these 2 samples. These blood samples will be taken by a member of the healthcare staff qualified to perform this type of procedure. If the results obtained with the 2 initial samples would be of interest to the Sponsor, the patient will be asked to come back for additional samplings with a maximum of 6 additional blood draws. The total volume of blood that will be taken over a 6 months period cannot exceed 500 milliliters with a maximum of 200 milliliters over a 30-day period for patients with a weight of min 50kg. The study has no other constraint.

The list of analysis planned to be performed on blood samples are presented below:

* Identification of the class II HLA antigens of each patient
* Study of the binding to HLA antigens of synthetic peptides
* Identification of peptides which, after binding to the HLA antigens, might induce a cytolytic response directed against the immune cells involved in the maintenance and triggering of the disease (i.e. non-cytolytic T cells recognising the same epitopes and APC presenting the same epitopes)
* Non selective genomic analysis (SNPs) in the scope of the single cell transcriptomic analysis technics

ELIGIBILITY:
Inclusion Criteria:

* Men or women, 18 to 65 years of age
* Patients with a confirmed diagnosis of Neuromyelitis Optica spectrum disorders according to IPND criteria (2015) and presenting a stabilized disease (no relapse) for at least 6 months.
* Patient positive for antibodies to human aquaporin 4
* Patients having granted their written informed consent to take part in this study

Exclusion Criteria:

* Ongoing pregnancy
* Ongoing treatment with immunosuppressive agents other than those listed below under section "authorized background therapy"
* Any investigational product in the last 3 months or less than 5 times the estimated half-life of the investigational product whichever is the longer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Measure in vitro binding of Imotopes® | Through study completion, an average of 1 year
  Characterize, in vitro, the binding of different Imotopes® to class II HLA antigens on PBMC isolated from patients with NMO
Measure Cytolytic response against Antigen-Presenting Cells (APC) | Through study completion, an average of 1 year
  Measure the ability of Imotopes® to generate a cytolytic response directed against the immune cells involved in the maintenance and triggering of the disease (i.e. non-cytolytic T cells recognising the same epitopes and APC presenting the same epitopes)

CONTACTS AND LOCATIONS:
Overall Officials: Jerome De Seze, MD, Principal Investigator — Hôpital de Hautepierre, Strasbourg
Locations (2):
- France (2):
  - Hôpital Pierre Wertheimer, Bron
  - Hôpital de Hautepierre, Strasbourg

IPD SHARING:
Plan to Share IPD: No